CLINICAL TRIAL: NCT03061305
Title: An Observational Trial Assessing the Clinical Benefit of Molecular Profiling in Patients With Solid Tumors
Brief Title: Assessing the Clinical Benefit of Molecular Profiling in Patients With Solid Tumors
Status: Terminated | Type: Observational
Why Stopped: Sponsor's discretion to termination due to business decision.
Sponsor: Strata Oncology (Industry)
Responsible Party: Sponsor
Other Study IDs: STR-001-001
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Adult Solid Tumor; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Neoplasms; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — leftover tumor tissue, DNA, RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many patients are treated for advanced cancer without knowledge of underlying molecular features that might indicate FDA approved therapies or potential eligibility for biomarker-selected clinical trials.

The Strata Trial (STR-001-001) has been initiated by Strata Oncology to evaluate the clinical benefit of systematic comprehensive genomic profiling for participants with advanced cancer using real-world data and endpoints, while assessing the proportion of participants available for clinical trials and approved targeted therapies in advanced and/or aggressive cancers. The Strata Trial uses surplus, or leftover, tumor specimens for molecular profiling and does not require additional study-specific procedures.

DETAILED DESCRIPTION:
Participants enrolled on the Strata Trial will submit surplus, clinical formalin-fixed paraffin-embedded (FFPE) tumor specimens for molecular profiling and a test report will be provided back to the investigator. For those participants identified as having molecular alterations associated with a Strata-affiliated therapeutic clinical trial and/or approved targeted therapy or trials, the Strata reports will provide additional relevant information.

All molecular profiling will be performed in the Strata Oncology CAP-accredited and CLIA-certified laboratory (Ann Arbor, MI). The molecular profiling assays will include tumor-only comprehensive genomic profiling (CGP) by next generation sequencing (NGS) of DNA and RNA covering a range of actionable genomic alterations, such as mutations (e.g. those in EGFR and BRAF), copy number alterations (e.g. ERBB2 amplifications), gene expression, gene fusions (e.g. ALK fusions), tumor mutation burden (TMB) and microsatellite instability status, and may include additional integrative DNA and RNA tests over time.

Participants may be followed for treatment changes and survival for three years from the time of enrollment and/or signed informed consent.

Participants may also be eligible for the Strata Trial Sub-Study at applicable Strata Trial sites. This sub-study is a sample collection study to support the development and evaluation of biomarker assays for patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 18 years of age.
* Subjects must have histologically documented solid tumors (including lymphoma and multiple myeloma).
* Specific criteria for individual tumor types are as follows:

  1. Participants with gliomas are eligible at any stage of disease
  2. Participants with pancreatic carcinoma are eligible at any stage of disease
  3. Participants with rare tumors (i.e. cancer started in an unusual place in the body, it is unusual type and requires special treatment) are eligible at stages II-IV.
  4. Participants with other tumor types must have recurrent, relapsed, refractory, metastatic, or advanced stages III or IV cancer.
  5. Participants with other tumor types must have recurrent, relapsed, refractory, metastatic, or advanced stages III or IV cancer.
* Must have an adequate formalin-fixed paraffin-embedded tumor specimen for genomic sequencing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with histologically-documented solid tumors (including lymphoma or multiple myeloma), that have surplus clinical FFPE tumor tissue (e.g. biopsy, fine needle aspiration, fluid cytology, surgical resection) will be eligible for the Strata trial.
Sampling Method: Non-Probability Sample
Enrollment: 58213 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Time to Treatment Discontinuation (TTD) | 3 years
  To evaluate TTD for participants who received an anticancer biomarker-guided therapy and, when available, as compared to prior TTD from prior anti-cancer therapy
Time to Next Treatment (TTNT) | 3 years
  To evaluate TTNT for participants who received and anticancer biomarker guided therapy and, when available, as compared to prior TTNT from prior anti-cancer therapy

SECONDARY OUTCOMES:
biomarker profiles indicative of potential clinical benefit and affiliate trial enrollment | 3 years
  To evaluate the proportion of participants with actionable genomic profiles that indicate a potential clinical benefit from standard of care biomarker-guided therapies or a clinical trial, and the proportion of participants who enroll on a clinical trial.
Correlation between real world endpoints and overall survival endpoint | 3 years
  To assess the correlation between real world endpoints and overall survival endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tomlins, MD, Study Director — Strata Oncology
Locations (40):
- United States (40):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Kaiser Permanente - Southern California, Pasadena, California
  - Kaiser Permanente - Northern California, Vallejo, California
  - SCL Health, Broomfield, Colorado
  - Kaiser Permanente Colorado, Denver, Colorado
  - Christiana Care Health System, Newark, Delaware
  - SwedishAmerican, Rockford, Illinois
  - Baptist Health, Lexington, Kentucky
  - Christus Health, Lake Charles, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Kaiser Permanente - Mid-Atlantic, Rockville, Maryland
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Minnesota Oncology - Coon Rapids, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Minnesota Oncology - Maplewood Cancer Center, Maplewood, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Metro-Minnesota Community Oncology Research Consortium, Minneapolis, Minnesota
  - Regions Hospital, Minneapolis, Minnesota
  - Minnesota Oncology - Minneapolis, Minneapolis, Minnesota
  - North Memorial Health Care, Robbinsdale, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Minnesota Oncology - Edina, Saint Louis Park, Minnesota
  - Minnesota Oncology - Woodbury Clinic, Woodbury, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - UNC REX Healthcare, Raleigh, North Carolina
  - Kettering Health Network, Kettering, Ohio
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Bon Secours St. Francis, Greenville, South Carolina
  - UTHealth - Memorial Hemann Cancer Institute, Houston, Texas
  - Bon Secours Midlothian, Midlothian, Virginia
  - MultiCare, Tacoma, Washington
  - Gundersen Health System, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Research Institute, Milwaukee, Wisconsin
  - ProHealth Care, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomlins SA, Hovelson DH, Suga JM, Anderson DM, Koh HA, Dees EC, McNulty B, Burkard ME, Guarino M, Khatri J, Safa MM, Matrana MR, Yang ES, Menter AR, Parsons BM, Slim JN, Thompson MA, Hwang L, Edenfield WJ, Nair S, Onitilo A, Siegel R, Miller A, Wassenaar T, Irvin WJ, Schulz W, Padmanabhan A, Harish V, Gonzalez A, Mansoor AH, Kellum A, Harms P, Drewery S, Falkner J, Fischer A, Hipp J, Kwiatkowski K, Lazo de la Vega L, Mitchell K, Reeder T, Siddiqui J, Vakil H, Johnson DB, Rhodes DR. Real-World Performance of a Comprehensive Genomic Profiling Test Optimized for Small Tumor Samples. JCO Precis Oncol. 2021 Aug 19;5:PO.20.00472. doi: 10.1200/PO.20.00472. eCollection 2021 Aug. PMID 34476329